CLINICAL TRIAL: NCT00534716
Title: Cannabis and Doping - Pharmacokinetics of Smoked Cannabis Under Controlled Clinical Conditions
Brief Title: Cannabis Cigarettes Used for Doping: Delta-9-Tetrahydrocannabinol (THC) Urine Detection
Status: Completed | Type: Observational
Sponsor: Federal Office of Sports, Switzerland (Other Government)
Responsible Party: Matthias Kamber, PhD, Federal Office of Sports, Office for Doping Control
Other Study IDs: KEK-33/07
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Cannabis; doping; THC; GC/MS; Pharmacokinetics; Volunteers
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study on volunteers is whether THC and short-living metabolites are suited to detect recent Cannabis smoking within urine doping control.

DETAILED DESCRIPTION:
About half of all positive doping cases in Switzerland have been related to Cannabis consumption (mainly recreational smoking). So far, the target analyte in urine is 11-nor-9-carboxy-THC (THC-COOH), the main metabolite of delta-9-tetrahydrocannabinol (THC), which is excreted up to several days after single use. However, the wide detection window of THC-COOH does not allow a conclusion concerning the impact on the physical performance. Therefore, the evaluation of other target analytes with shorter elimination half-lives is needed and the aim (primary endpoints) of the present study. This pharmacokinetic, open, 1-session trial on 12 healthy, male, infrequently Cannabis smoking volunteers is focussed on the GC/MS profiling of THC and metabolites in urine and plasma after standardized smoking of a single 7% THC Cannabis cigarette of the Dutch Ministry of Health, Welfare & Sport, Office of Medicinal Cannabis. Pharmacodynamic measurements (secondary endpoints) include the side-effects monitoring by using Visual Analog Scales and checking vital functions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects; light (max. 1/month), infrequent Cannabis smokers, medium (max. 15/month) tobacco smokers experienced in the inhalation technique; age 20-30 years; body weight 75+/-15 kg; evaluation based on normal medical history, physical examination, laboratory tests (safety lab), normal lung functions (spirometry).
* Informed consent after information (written) by the study physician and principal investigator on nature, significance and scope of the trial.
* Informed consent by the volunteer regarding transmitting trial-related data to the sponsor and to the competent control authorities.

Exclusion Criteria:

* Hypersensitivity to cannabinoids. - Regular (more than once per month, weekly or daily) Cannabis use. - The use of alcohol, any medication or drugs, especially Cannabis, within the last 2 days prior to and during the 1-day session is not allowed. Cannabis use is also not allowed during the following 11 days of urine collection, i.e. up to the end of the study.
* Positive Cannabis urine test before the session.
* Driving any vehicle, and operating with machines during and within 48 h after the session.
* Psychotic or vulnerable subjects.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male subjects; light (max. 1/month), infrequent Cannabis smokers, medium (max. 15/month) tobacco smokers experienced in the inhalation technique; age 20-30 years; body weight 75+/-15 kg, normal medical history physical examination, passed laboratory tests (safety lab), normal lung functions (spirometry).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Brenneisen, PhD, Prof, Principal Investigator — University of Bern, Dept. Clinical Research
Locations (1):
- Clinical Investigation Unit (CIU), University Hospital ("Inselspital"), Bern, Switzerland